CLINICAL TRIAL: NCT00044915
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetic / Pharmacodynamic Effects of a Targeted Exposure of Intravenous Repinotan in Patients With Acute Ischemic Stroke
Brief Title: Repinotan in Patients With Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer HealthCare AG
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100282
Record Dates: First submitted 2002-09-06; First posted 2002-09-09 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Stroke; Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke Without Hemorrhage
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: Repinotan HCl (BAYX3702)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Repinotan HCl (BAYX3702) — All patients receive 1.25 mg of repinotan
  Arms: Arm 1
Drug: Placebo — All patients receive 1.25 mg of placebo
  Arms: Arm 2

SUMMARY:
The purpose of this trial is to evaluate Repinotan HCl in patients with acute ischemic stroke. At study entry patients will be randomized to Repinotan HCl or placebo in a 1:1 ratio. The total treatment period wil be 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke of hemispheric localization (exclude brainstem and cerebellum), of suspected thromboembolic origin.
* Males or females aged 18 years or over.
* National Institute of Health Stroke Scale (NIH-SS) total score 8 to 23 with a motor deficit >/= 2 (for either one arm or leg) and level of consciousness < 2 and at least one of the following: Visual field deficit, neglect, or aphasia. If a patient receives t-PA, NIH-SS must be performed prior to receiving the study drug but after infusion of t-PA is initiated.
* Signed informed consent from patient or legally authorized representative

Exclusion Criteria:

* CT scan evidence of:
* Clearly defined areas of hypodensity indicating infarction of >1/3 of the MCA territory or evidence of significant mass effect with shift of midline or major areas of sulcal effacement associated with loss of cortical definition (grey-white distinction). Minor early CT changes are common in MCA strokes and patients with early or subtle changes are eligible.
* A primary intra-cerebral haemorrhage or any finding not consistent with an acute ischemic stroke as the cause of presenting symptoms.
* Clinical evidence of acute stroke due to lacunar infarct (pure motor hemiplegia; pure sensory deficit, ataxia/clumsy hand syndromes)
* Neurological (other than the presenting stroke) or psychiatric conditions that may affect the patient's functional status and/or that may interfere with the patient's assessment
* Clinically relevant pre-existing neurological deficit (Historical Rankin score >/= 2 regardless of cause)
* Generalized seizures having developed since the onset of stroke symptoms
* Systolic blood pressure > 210 or < 110 mmHg (confirmed by up to three readings prior to randomization)
* Diastolic blood pressure > 110 or < 60 mmHg (confirmed by up to three readings prior to randomization)
* Myocardial infarction within 3 months, unstable angina within 3-5 days prior to starting infusion, unstable supra-ventricular and/or ventricular arrhythmia, severe conduction defect (AV block grades 2 and 3), complete left or right Bundle Branch Block, bradycardia (heart rate [HR] less than 50 bpm), uncompensated heart failure
* History of myocarditis, cardiomyopathy or aortic stenosis
* Patients known to have prolonged QTc intervals (inherited and sporadic syndromes of QTc prolongation or QTc interval > 450 msec males and 470 msec females on baseline ECG) or using Class IA or Class III antiarrhythmic drugs (e.g., quinidine, procainamide, amiodarone, sotalol)
* Any patients that require initiation of new digoxin therapy are excluded. Patients already on digoxin therapy (for at least 1 month stable dose) at time of enrollment will be allowed in the study.
* Electrolyte imbalance at baseline. Should the results not be available before starting the study drug infusion, the patients will be allowed in the study providing that the corrective therapy of any abnormal electrolyte results is implemented immediately upon availability of the laboratory report.
* Any conditions predisposing to electrolyte imbalances (e.g., chronic vomiting, anorexia nervosa, bulimia nervosa) will also be excluded at baseline.
* Participation in a research protocol for investigation of a pharmaceutical agent or innovative invasive procedure (including intra-arterial t-PA) within the past 30 days
* Previously in the BRAIN-Study or treated with repinotan
* Life expectancy of less than 6 months due to comorbid conditions
* Any other known clinically significant medical disorder (e.g., cardiovascular, gastrointestinal, hepatic, renal, endocrine, major uncompensated metabolic disturbances, respiratory, immunological, hematological or bleeding disorder, cancer, AIDS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 782 (Actual)
Dates: Start 2000-12; Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (112):
- United States (28):
  - Los Angeles, California
  - Oceanside, California
  - San Diego, California
  - San Jose, California
  - Boynton Beach, Florida
  - Fort Lauderdale, Florida
  - Ocala, Florida
  - Tampa, Florida
  - Decatur, Georgia
  - Honolulu, Hawaii
  - Des Moines, Iowa
  - Baltimore, Maryland
  - Robbinsdale, Minnesota
  - Great Falls, Montana
  - Edison, New Jersey
  - Ridgewood, New Jersey
  - New Hyde Park, New York
  - Stony Brook, New York
  - Chapel Hill, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Upland, Pennsylvania
  - Beaufort, South Carolina
  - Chattanooga, Tennessee
  - Houston, Texas
  - Bellevue, Washington
- Australia (5):
  - Gosford, New South Wales
  - New Lambton Heights, New South Wales
  - Southport, Queensland
  - Hobart, Tasmania
  - Melbourne, Victoria
- Austria (3):
  - Klosterneuburg, Lower Austria
  - Linz, Upper Austria
  - Vienna, Vienna
- Belgium (2):
  - Bornem
  - Bruxelles - Brussel
- Canada (18):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Lethbridge, Alberta
  - North Vancouver, British Columbia
  - Penticton, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Saint John, New Brunswick
  - Halifax, Nova Scotia
  - London, Ontario
  - Mississauga, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Greenfield Park, Quebec
  - Québec, Quebec
  - Saskatoon, Saskatchewan
- Finland (4):
  - Helsinki
  - Kuopio
  - Lahti
  - Mikkeli
- France (2):
  - Bordeaux
  - Nice
- Germany (20):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Aschaffenburg, Bavaria
  - Bad Neustadt an der Saale, Bavaria
  - Erlangen, Bavaria
  - München, Bavaria
  - Nuremberg, Bavaria
  - Regensburg, Bavaria
  - Würzburg, Bavaria
  - Frankfurt am Main, Hesse
  - Greifswald, Mecklenburg-Vorpommern
  - Cologne, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Minden, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Kaiserslautern, Rhineland-Palatinate
  - Leipzig, Saxony
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
- Miskolc, Hungary
- Israel (7):
  - Petah Tikva, Isarel
  - Ashkelon
  - Haifa
  - Holon
  - Nahariya
  - Tel Aviv
  - Tel Litwinsky
- Italy (10):
  - Como
  - L’Aquila
  - Milan
  - Pavia
  - Perugia
  - Reggio Emilia
  - Roma
  - Verona
  - Vibo Valentia
  - Vicenza
- Netherlands (2):
  - Groningen
  - Nijmegen
- Spain (5):
  - Santiago de Compostela, A Coruña
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Valencia, Valencia
  - Zaragoza, Zaragoza
- Sweden (2):
  - Stockholm
  - Umeå
- United Kingdom (3):
  - Leicester, Leicestershire
  - Glasgow, Strathclyde
  - Dundee, Tayside